CLINICAL TRIAL: NCT05127876
Title: Ephedrine Versus Ondansetron in the Prevention of Hypotension During Cesarean Delivery: a Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Ephedrine Versus Ondansetron During Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raham Hasan Mostafa, MD, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R 04 2022
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Spinal Induced Hypotension
Keywords: cesarean section; Bezold-Jarisch reflex; ondansetron
MeSH Terms: interventions — Ondansetron; Ephedrine; Saline Solution

STUDY DESIGN:
Intervention Model Description: According to patients' randomized groups, study medication was given over 1 min, 5 min before spinal anesthesia
  Patients were randomly assigned into 1 of 4 groups, using computer generated sequence and opaque envelopes, according to the prophylactic intravenous drug dose used:
  * Group E: were administered intravenous ephedrine 10 mg diluted in 10 mL 0.9% saline over 1 minute;
  * Group OL: were administered intravenous ondansetron 4 mg diluted in 10 mL 0.9% saline over 1 minute;
  * Group OH: were administered intravenous ondansetron 8 mg diluted in 10 mL 0.9% saline over 1 minute;
  * Group P: was a control group who received 0.9% saline 10 mL over 1 minute as a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study at the level of patients, careproviders, and outcome assessors. Anesthesiologists, surgeons, and operating personnel did not know which study treatment was used. Syringes were identical in terms of volume, color, viscosity, and odor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group E (Experimental): Monitoring with pulse oximetry, noninvasive blood pressure measurement and electrocardiogram was established on arrival to the operating room Group E: were administered intravenous ephedrine 10 mg diluted in 10 mL 0.9% saline over 1 minute; Then under aseptic precautions, spinal anesthesia was administered.
  Interventions: Drug: EPHEDrine 10 Mg/mL-NaCl 0.9% Intravenous Solution
- Group OL (Experimental): Monitoring with pulse oximetry, noninvasive blood pressure measurement and electrocardiogram was established on arrival to the operating room Group OL: were administered intravenous ondansetron 4 mg diluted in 10 mL 0.9% saline over 1 minute; Then under aseptic precautions, spinal anesthesia was administered.
  Interventions: Drug: Ondansetron 4 MG
- Group OH (Experimental): Monitoring with pulse oximetry, noninvasive blood pressure measurement and electrocardiogram was established on arrival to the operating room Group OH: were administered intravenous ondansetron 8 mg diluted in 10 mL 0.9% saline over 1 minute; Then under aseptic precautions, spinal anesthesia was administered.
  Interventions: Drug: Ondansetron 8mg
- Group P (Placebo Comparator): Monitoring with pulse oximetry, noninvasive blood pressure measurement and electrocardiogram was established on arrival to the operating room Group P: was a control group who received 0.9% saline 10 mL over 1 minute as a placebo.
  Then under aseptic precautions, spinal anesthesia was administered.
  Interventions: Other: 10 mL normal saline

INTERVENTIONS:
Drug: Ondansetron 4 MG — Ondansetron 4mg was given over 1 min, 5 min before spinal anesthesia
  Other Names: Low dose ondansetron group
  Arms: Group OL
Drug: Ondansetron 8mg — Ondansetron 8mg was given over 1 min, 5 min before spinal anesthesia
  Other Names: Higher dose Ondanseteron group
  Arms: Group OH
Drug: EPHEDrine 10 Mg/mL-NaCl 0.9% Intravenous Solution — Ephedrine 10mg was given over 1 min, 5 min before spinal anesthesia
  Other Names: Ephedrine group
  Arms: Group E
Other: 10 mL normal saline — 10 mL normal salinwe 0.9% was given over 1 min, 5 min before spinal anesthesia
  Other Names: Placebo group
  Arms: Group P

SUMMARY:
More than 30% of the patients receiving spinal anesthesia develop hypotension. Hypotension developed during cesarean section (C/S) under spinal anesthesia may jeopardize uteroplacental circulation leading to fetal compromise and even fetal death.

The effect of prophylactic ondansetron on blood pressure after spinal anesthesia has not been compared in a clinical trial with that of a vasoconstrictor. The investigators will compare ephedrine and ondansetron for the prevention of maternal hypotension after spinal anesthesia for elective cesarean delivery.

DETAILED DESCRIPTION:
Some vasopressive drugs including ephedrine and phenylephrine have been widely used to prevent maternal hypotension. Although ephedrine has mixed a-adrenoceptor activity , it maintains arterial pressure mainly by increases in cardiac output and heart rate as a result of its predominant activity on β1-adrenoceptors. It has been demonstrated that ondansetron preloading with crystalloid infusion reduces maternal hypotension in parturient women undergoing cesarean delivery.

Ondansetron has been widely used in the clinic to prevent nausea and vomiting caused by cancer chemotherapy, radiation therapy, and surgery. Ondansetron has been proven as a well-tolerated drug, but the most common side effects of ondansetron include headache, constipation, diarrhea, asthenia, and somnolence.

ELIGIBILITY:
Inclusion Criteria:

* age >18, <40 years;
* American Society of Anesthesiologists physical status I or II;
* term pregnancy
* singleton pregnancy;
* elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Patients with a history of diabetes mellitus other than gestational diabetes,
* hypertension,
* body mass index >40 kg/m2,
* complicated pregnancy, allergy to study drugs,
* long QT syndrome,
* Contraindication to spinal anesthesia
* Patients who required general anesthesia were withdrawn from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 168 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Maternal hypotension | 45 minutes
  Mean arterial blood pressure was recorded every 2 minute for 10 minutes then every 5 minutes until delivery. Time of intrathecal injection was considered as 0 min.

SECONDARY OUTCOMES:
Apgar score | 5 min after fetal delivery
  1and 5 min after fetal delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request